CLINICAL TRIAL: NCT07016906
Title: MRI Assessment of Knee Kinematics From Extension to Flexion - Exploratory Study
Acronym: FLEXIGEN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A00579-40
Record Dates: First submitted 2025-06-03; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI arm (Experimental): Knee MRI at different degrees of flexion
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Knee MRI at different degrees of flexion

SUMMARY:
During flexion of the knee, internal rotation of the tibia associated with translation of the tibial plateaus in relation to the femoral condyles is automatically induced. This mechanism combines a sliding phenomenon and a rolling phenomenon of the condyles on the plate, the latter being known as 'roll-back'. In 2024, imaging analyses of the knee, and in particular MRI, are carried out with the leg in extension.

MRI of the knee at different degrees of flexion would enable to assess the sliding and roll-back phenomena, in order to gain a better understanding of knee kinematics.

However, MRI of the knee at different degrees of flexion is limited by the size of the MRI machines and especially by the knee antennae, which are narrow and do not allow flexion beyond 30°. In this context, the only solution for carrying out an MRI study on knees in flexion would be to carry out this examination with an antenna that allows the knee to be positioned at different angles of flexion. This particular type of antenna only exists in veterinary schools, where they are used in particular for horses.

Consequently, this study is based on the assumption that the kinematics of the knee can be assessed using MRI with an antenna for veterinary use.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (no damage to either knee)
* Male or female, aged between 18 and 40
* Healthy volunteer affiliated to or benefiting from a social security scheme
* A healthy French-speaking volunteer who has signed an informed consent form.

Exclusion Criteria:

* Contraindication to MRI
* Joint osteoarthritis
* BMI > 30
* Previous trauma or surgery to the knee
* Recurrence of sprains
* Knee trauma other than sprain
* Protected person: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.
* Pregnant or breast-feeding woman

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
femorotibial knee kinematics | Day 1
  The kinematics of the knee will be described on the basis the femorotibial contact surfaces at the level of the medial tibial plateau and the lateral tibial plateau at each degree of flexion, during an MRI acquisition. Contact surfaces will be measured in mm2.

CONTACTS AND LOCATIONS:
Locations (1):
- Hawkcell, Marcy-l'Étoile, France

IPD SHARING:
Plan to Share IPD: No